CLINICAL TRIAL: NCT04258176
Title: A Multidisciplinary Outpatient Pathway
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 634802
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Multimorbidity
Keywords: outpatient; multimorbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Patients seen in the multidisciplinary pathway
  Interventions: Other: Multidisciplinary outpatient pathway
- Comparison group: Multimorbid patients seen several outpatient clinics who did not undergo the trajectory

INTERVENTIONS:
Other: Multidisciplinary outpatient pathway — Coordinators, assigned to improve the care flow, review and align the patient's appointments and tests in agreement with the patient's wishes. Outpatient consultations are arranged to take place the same day and schedules for care providers are coordinated. The patients' attendance in outpatient clinics are planned sequentially where the delivering specialty writes a summary to the subsequent specialty. Afterwards, the involved physicians and nurses attend an interdisciplinary conference, resulting in a joint treatment plan, with feedback and notice of modifications, which is delivered to the patient and general practice.
  Groups: Intervention group

SUMMARY:
Patients with complex chronic multiple illnesses constitute an increasing challenge and more evidence-based knowledge of effective practice is required. In Denmark and the rest of the world, improved health care, public health, and increased focus on early diagnosis have led to increases in life expectancy resulting in a growing population of older people living with multiple long-term conditions (multimorbidity). Today, every fourth Dane suffers from more than one concomitant chronic or severe disease, estimated to rise to 60% for those over 65 years.

National and international health care is organised and targeted as specialised, mono-diagnostic efforts for single diseases leading to lack of coordination and failure to integrate multidisciplinary patient trajectories. Danish research shows that general practice is challenged by insufficient collaboration between professionals involved in the treatment. Despite this, there exists limited evidence of initiatives aiming to improve care for multimorbid patients.

This study aims to:

1. identify chronic multimorbid patients and to analyse their use of two or more outpatient clinics, their general use of health care utilisations and their disease pattern and characteristics (Cross-sectional study using national registers).
2. develop an innovative organisational structure around a multidisciplinary outpatient pathway for multimorbid patients and to pilot-test it (feasibility study)
3. phase-III test a multidisciplinary outpatient pathway and to preliminarily evaluate the effects in patients and health professionals and on resource utilisations (effect study)

DETAILED DESCRIPTION:
Background Patients with complex chronic multiple illnesses constitute an increasing challenge and more evidence-based knowledge of effective practice is required. In Denmark and the rest of the world, improved health care, public health, and increased focus on early diagnosis have led to increases in life expectancy resulting in a growing population of older people living with multiple long-term conditions (multimorbidity). Today, every fourth Dane suffers from more than one concomitant chronic or severe disease, estimated to rise to 60% for those over 65 years. Multimorbidity is more prevalent in women, rises with declining social status and is associated with poorer quality-of-life. With an increasing proportion of multimorbid patients, the prevalence of polypharmacy will increase. A multisymptomatic and complicated disease pattern applies to both physical and mental illness, multiplicative effects can create a need for people within different specialities working together. Earlier studies show, that the most common chronic diseases are diabetes, cardiovascular disease, cancer, chronic obstructive pulmonary disease and asthma. Comorbid diseases tend to compound and interact, for example, COPD and diabetes are often seen in combination with cardiovascular disease.

Everyday-life of multimorbid patients is influenced by drug consumption, frequent visits to general practice, hospitalisations and outpatient clinics. A recent study showed that patients with three chronic conditions visit health professionals five times a month and spend 50-71 hours per month on health-related activities. However, studies on derivative effects of multimorbidity are scarce and research focus is primarily placed on mainly health services. Multimorbid patients experience and are in reality exposed to lack of coordination, lack of inter-disciplinary communication and overall poor care management. Individual resources and priorities in everyday life play a dominant role in navigating the tension between everyday life and the health care system. This is often extremely demanding for patients to navigate in.

National and international health care is organised and targeted as specialised, mono-diagnostic efforts for single diseases leading to lack of coordination and failure to integrate multidisciplinary patient trajectories. Danish research shows that general practice is challenged by insufficient collaboration between professionals involved in the treatment. Despite this, there exists limited evidence of initiatives aiming to improve care for multimorbid patients. Previous initiatives involve getting patients to take more active part in their disease, creating disease insight, involving case managers, patient-shared medical appointments, collaborative models and communication technology. Present on-going studies focusing on interventions for multimorbid patients are also few.

In conclusion, the evidence is sparse on collaborative approaches directed at multimorbid patients and on organising health care systems to accommodate this.

Objectives and hypotheses Hypothesis 1 Multimorbid patients have numerous contacts to outpatient clinics and are characterised as being older patients with common chronic diseases, a complicated disease pattern and frequent users of health care utilisations.

Objective 1: To identify chronic multimorbid patients and to analyse their use of two or more outpatient clinics, their general use of health care utilisations and their disease pattern and characteristics.

Hypothesis 2: It is feasible to convert several outpatient clinic pathways to one multidisciplinary outpatient pathway and to structure an organisation around it.

Objective 2: To develop an innovative organisational structure around a multidisciplinary outpatient pathway for multimorbid patients and to pilot-test it.

Hypothesis 3: Patients and health care professionals find it advantageous to convert outpatient visits for multimorbid patients to a multidisciplinary outpatient pathway, and the use of resources will lower.

Objective 3: To phase-III test a multidisciplinary outpatient pathway and to preliminarily evaluate the effects in patients and health professionals and on resource utilisations.

Materials and Methods

Objective 1:

In a national cross-sectional study, data on multimorbid patients is obtained using validated Danish registries, processed with remote access to Statistics Denmark.

Inclusion criteria:

* Patients who are diagnosed with more than one chronic disease
* Seen in more than one outpatient clinic (within 18 months, 12 months, 6 months, 3 months)
* ≥18 years of age.

Exposure and outcomes: Primary exposure constitutes chronic diseases occurring in multimorbid patients with classification a priori. Based on diagnoses (selected diagnoses chosen from previous studies), clinical, socio-demographic characteristics and the need for health care are investigated. We wish to demonstrate how these exposures are distributed by the number of concomitant outpatient visits within different time intervals of 18 months, 12 months, 6 months, 3 months.

Objective 2:

In a feasibility-design efforts will be devoted to setting up an innovative multidisciplinary outpatient pathway based on recommendations for complex interventions in the health system. It involves the process of going from a conceptual to an operational setup.

Procedure: A multidisciplinary outpatient pathway will be established at the University Research Clinic for Innovative Patient Pathways. Through literature review and specialist opinions, interviews, the intervention will consist of two or more disciplines collaborating in establishing a treatment plan for the patient. A process manual of the individual phases and a participatory cooperative approach will be used. A steering group will involve plastic organic groups (health care professionals, patients, general practitioners), which will contribute along with the hospital's task force team (center management, senior health care professionals, representatives of quality development) through process support.

Exposure and outcomes: In the multidisciplinary outpatient pathway, health care professionals will collaborate between medical specialties and examinations gathered for one joint encounter with the patient. An integrated discharge summary is sent to general practice. The exact structure and composition of the multidisciplinary outpatient pathway is part of the feasibility study. Interviews are conducted on patients and healthcare professionals to assess their experience with the pathway. Also a process evaluation is made.

Study 3: To phase-III test a multidisciplinary outpatient pathway and to preliminary evaluate the effects in patients and healthcare professionals and on resource utilisations.

In a prospective study with difference-in-difference analysis, a cohort of multimorbid patients seen in outpatient clinics is included based on the composition from the feasibility study.

Exposure: The newly established multidisciplinary outpatient pathway. Outcomes: In paired measurements, Patient Reported Experience Measures (PREM) are recorded in questionnaires before and after trajectories in conventional mono-disciplinary outpatient clinics are converted to trajectories in the multidisciplinary outpatient pathway. Questionnaires are compiled according to the literature of existing, validated questionnaires and supplemented by ad hoc questions when no existing questionnaire exists). Questionnaires are set up in the processing program, REDCap and sent through "e-boks" merged with doc2mail where replies are entered directly in REDCap through a link. Questionnaires will also be sent by letter.

The cohort will be followed for one year for data collection on health care utilisations (e.g. admissions, visits to outpatient clinics, redeemed prescriptions, contacts to general practice or emergency medical services, hospital activity/examinations). A control group of patients from other hospitals with trajectories in outpatient clinics are matched by gender, age, disease, comorbidity, and length of disease. Difference-in-difference comparisons are made on healthcare utilizations one year prior to the index date (first consultation with the new pathway). Data is retrieved from national registers.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen on two or more outpatient Clinics at Silkeborg Regional Hospital
* 18 years old or older
* Specialties involved: Nephrology, rheumatology, cardiology, endocrinology, pulmonology
* Listed for future appointments in two or more outpatient clinics
* Days between appointments less than 43

Exclusion Criteria:

* Patients only undergoing patient education
* Appointments in relation to science or diagnosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multimorbid patients who have several trajectories and appointments in outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
PREM - PACIC | August 2018 - August 2020 (approximately)
  Patient reported outcome measures: questionaires incl. The Patient Assessment of Chronic Illness Care (PACIC). This is a 20-item scale with a 5-point scale from (1(never) to 5 (allways). PACIC is reported as an avarage of the 20 items.
PREM - MTBQ | August 2018 - August 2020 (approximately)
  Patient reported outcome measures: questionaires incl. The Multimorbidity Treatment Burden Questionnaire. This is a 10-item scale with a 6-point scale. The Multimorbidity Treatment Burden Questionnaire (MTBQ) questionnaire is designed to measure treatment burden (the effort of looking after one's health) in patients with multimorbidity (multiple long term conditions). You calculate the average score from the questions answered. Multiple the average score by 25 to give a global MTBQ score from 0-100
Attendance in outpatient clinics | August 2018 - August 2021 (approximately)
  Number of times patients are coming to the hospital for outpatient visits

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, Study Director — Diagnostic Center, University Research Clinic for Innovative Patient Pathways
Locations (1):
- University Research Clinic for Innovative Patient Pathways, Diagnostic Centre, Silkeborg Regional Hospital, Silkeborg, Central Jutland, Denmark